CLINICAL TRIAL: NCT06616194
Title: AN INTERVENTIONAL, EFFICACY, AND SAFETY, PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY WITH AN OPEN-LABEL EXTENSION TO INVESTIGATE RIMEGEPANT IN MIGRAINE PREVENTION IN ADOLESCENTS 12 TO LESS THAN 18 YEARS OF AGE WITH CHRONIC MIGRAINE
Brief Title: A Study to Learn About the Study Medicine Called Rimegepant in Adolescents With Frequent Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4951013; BHV3000-320 (Other: Alias Study Number); 2023-505601-16-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Chronic migraine; adolescents; rimegepant,; cgrp
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rimegepant (Experimental): Experimental medicine under study
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator): A placebo does not have any medicine in it but looks just like the medicine being studied.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75 mg orally disintegrating tablets
  Arms: Rimegepant
Drug: Placebo — Matching placebo oral disintegrating tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the effect of a study medicine called rimegepant in adolescents who have frequent migraine attacks.

Rimegepant is a tablet that dissolves when you put it on or under your tongue.

The study will enroll participants who have headache for 15 days (or more) every month, of which 8 days (or more) of migraine every month, and each untreated attack lasts for an average of 4-72 hours

In the 1st part of the study approximately half of the participants will receive a rimegepant tablet every other day, and approximately half of the participants will receive an inactive oral tablet (that looks the same as the rimegepant tablet) every other day.

Participant experiences when they are taking the study medicine will be compared to when they are taking the inactive tablet. This will help to determine if the study medicine is safe and effective. The 1st phase of the study will last 3 months.

In the 2nd part of the study all the participants who stay on study will receive rimegepant tablet every other day. This 2nd phase of the study will last 1 year. This will help determine if the study medicine is safe when taken for a long period.

Those who will participate in both phases will have up to 19 visits at the study clinic, about one every 4 weeks (this may vary from 2 to 8 weeks interval during the study). Home health visits may occur as well. A health check and blood sample will be conducted at all visits. Participants will have to complete a daily diary to record the migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* At least a 6 month history of migraine (with or without aura)
* 15 or more headache days/month
* 8 or more migraine days/month
* Migraine lasting 4-72 hours if untreated

Exclusion Criteria:

* Unrelenting headache
* Current psychiatric condition uncontrolled or untreated
* History of suicidal behavior or the subject is at risk of self-harm
* History of alcohol abuse and/or illicit drug use
* History of severe drug allergy
* Use of more than one medication for migraine prevention/prophylaxis
* Participation in another clinical trial at the same time

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
Number of migraine days per month | 12 Weeks
  Efficacy of rimegepant relative to placebo, measured as mean change from the baseline in the number of migraine days per month

SECONDARY OUTCOMES:
Efficacy of rimegepant relative to placebo measured as the mean change from baseline in the number of acute migraine-specific medication days per month | 12 Weeks
  Change in the use of acute migraine-specific medication days per month
Efficacy of rimegepant relative to placebo measured the mean change from baseline in the number of headache days per month | 12 Weeks
  Change in headache days per month
Efficacy of rimegepant relative to placebo measured as the percentage of participants with at least 50% reduction from baseline in number of moderate or severe migraine days per month | 12 weeks
  Change in moderate or severe migraine days per month
Efficacy of rimegepant relative to placebo measured as the mean change from baseline in the Pediatric Quality of Life (PedsQL™) total score | 12 Weeks
  Change in the Quality of Life
Efficacy of rimegepant relative to placebo measure as the mean change from baseline in the number of acute headache medication days per month, and acute migraine-specific medication days per month | 12 Weeks
  Change in headache and migraine rescue medication(s) used
Safety of rimegepant relative to placebo, and safety of rimegepant given for a long period of time measured as the number and percentage of participants with adverse event by severity and overall | Up to 15 months
  Safety and tolerability of the study drug
Safety of rimegepant relative to placebo, and safety of rimegepant given for long period of time measured as the number and percentage of participants with liver-related adverse event and action taken | Up to 15 Months
  Safety monitoring of adverse events of special interest
Efficacy of rimegepant relative to placebo measured as mean change from baseline in the PedMIDAS total score | 12 Weeks
  Change in the Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (106):
- United States (26):
  - Adult & Child Neurology Medical Associates, Long Beach, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Chicago Headache Center and Research Institute, Naperville, Illinois
  - New England Regional Headache Center, Worcester, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Clinvest Headlands Llc, Springfield, Missouri
  - Rutgers University, New Brunswick, New Jersey
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Duke Health Center Creekstone, Durham, North Carolina
  - Duke Lenox Baker Children's, Durham, North Carolina
  - Duke Children's Health Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center ( WFUBMC ), Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Avera Medical Group Pediatric Specialists, Sioux Falls, South Dakota
  - Avera Research Institute - Sioux Falls, Sioux Falls, South Dakota
  - Avera Medical Group Pediatrics - Dawley Farm, Sioux Falls, South Dakota
  - Dell Children's Medical Center, Austin, Texas
  - Headlands Research-El Paso, El Paso, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Granger Medical Holladay - Holladay Clinic, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (4):
  - University Of Alberta Hospital, Edmonton, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - CaRe Clinic, Red Deer, Alberta
  - London Health Sciences Centre - Verspeeten Family Cancer Centre, London, Ontario
- China (14):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Wuhan Children's Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shanghai Children's Hospital, Shanghai
  - The Second Affiliated Hospital of Hebei Medical University, Shijiazhuang
- Czechia (5):
  - Detska nemocnice FN Brno, Brno, Brno-město
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava, Moravskoslezský kraj
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice v Motole, Prague, Praha 5
- Finland (7):
  - Terveystalo Oulu, Oulu, North Ostrobothnia
  - Kuopion Yliopistollinen Sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - New Children's Hospital, Helsinki, Uusimaa
  - Terveystalo Tampere, Tampere
  - Terveystalo Pulssi, Turku
- Hungary (5):
  - Dr. Kenessey Albert Kórház, Balassagyarmat, Nógrád megye
  - Nagykanizsai Kanizsai Dorottya Korhaz, Nagykanizsa, Zala County
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- India (7):
  - Artemis hospital, Gurugram, Haryana
  - Fortis Memorial Research Institute, Gurugram, Haryana
  - Mallikatta Neuro Centre, Mangalore, Karnataka
  - JSS Hospital, Mysore, Karnataka
  - Chopda Medicare & Research Centre Pvt. Ltd; Magnum Heart Institute, Nashik, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
- Italy (8):
  - ASL1 Avezzano-Sulmona-L'Aquila, L’Aquila, Abruzzo
  - Ospedale San Paolo Bari, Bari, Apulia
  - AOU Policlinico Umberto I, Rome, Lazio
  - IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - Asst Spedali Civili Di Brescia, Brescia
  - I.C.O.T. Università La Sapienza, Latina
  - Fondazione Istituto Neurologico C. Mondino, Pavia
  - IRCCS San Raffaele Roma, Roma
- Japan (7):
  - Konan Medical Center, Kobe, Hyōgo
  - Yamaguchi Clinic, Nishinomiya, Hyōgo
  - Tominaga Clinic, Osaka, Osaka
  - Tokyo Headache Clinic, Shibuya-ku, Tokyo
  - Nagaseki Headache Clinic, Kai, Yamanashi
  - Tanaka Neurosurgery&Headache Clinic, Kagoshima
  - Tennoji Department of Neurosurgery, Osaka
- Poland (9):
  - AthleticoMed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny, Wroclaw, Lower Silesian Voivodeship
  - MedicArt Sp. z o. o., Wroclaw, Lower Silesian Voivodeship
  - NZOZ Neuromed M.i M. Nastaj, Lublin, Lublin Voivodeship
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin, Lublin Voivodeship
  - Dr Sękowska Leczenie Bólu, Warsaw, Masovian Voivodeship
  - Neurosphera, Warsaw, Masovian Voivodeship
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw, Masovian Voivodeship
- Slovakia (6):
  - Detska fakultna nemocnica s poliklinikou Banska Bystrica, Banská Bystrica
  - IN MEDIC s.r.o., Bardejov
  - Narodny ustav detskych chorob, Bratislava
  - Detsky neurolog s.r.o., Bratislava
  - KONZILIUM s.r.o., Dubnica nad Váhom
  - Univerzitna nemocnica Martin, Martin
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitario HM Puerta del Sur, Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - CHUVI- Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951013